CLINICAL TRIAL: NCT02290574
Title: Efficacy of Neoadjuvant Thermo-Radio-chemotherapy for Locally Advanced Rectal Cancer Before Laparoscopic Total Mesorectal Excision: Prospective Phase II Trial
Brief Title: Efficacy of NeoThermo-Radio-chemotherapy for LA Rectal Cancer Before Laparoscopic TME: Prospective Phase II Trial
Acronym: NEOTREAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Park Hee Chul, Assocate Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-10-019
Record Dates: First submitted 2014-11-06; First posted 2014-11-14 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Locally Advanced Rectal Cancer
MeSH Terms: interventions — Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thermo-radio-chemotherapy arm (Experimental): Hyperthermia with concurrent chemo-radiation therapy
  Interventions: Radiation: Hyperthermia with concurrent chemo-radiation therapy

INTERVENTIONS:
Radiation: Hyperthermia with concurrent chemo-radiation therapy

SUMMARY:
The investigators start this prospective study to evaluate the efficacy of laparoscopic total mesorectal excision after concurrent chemo-radiation therapy with hyperthermia in locally advanced rectal cancer.

DETAILED DESCRIPTION:
The current standard treatment of locally advanced rectal cancer is neoadjuvant concurrent chemo-radiation therapy (CCRT) followed by total mesorectal excision (TME). Recently, laparoscopic surgery is getting substitute open surgery based on the advantages of early recovery, short admission, less pain, less blood loss, and little scar without compromising oncologic outcomes.

It is reported that hyperthermia is effective in synthetic (S) phase, Low oxgen pressure, acidic, and low perfusion site which are known as radio-resistant. Because of these characteristics, it considered as the most valuable radiosensitizer in cancer treatment, theoretically. Furthermore, mild hyperthermia (41 to 41.5 ºC) can promote tumor reoxygenation.

Based on those background, the investigators start this prospective study to evaluate the efficacy of laparoscopic TME after CCRT with hyperthermia in locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 20 years or older
* pathologically confirmed rectal cancer
* Eastern Cooperative Oncology Group performance status 0 to 2
* Candidate of laparoscopic TME
* Optimal bone marrow function
* Locally advanced rectal cancer confirmed by magnetic resonance imaging

Exclusion Criteria:

* Extrapelvic metastasis
* Previous pelvic irradiation
* Current status of pregnant or breast feeding
* Confirmed other malignancy within two years except thyroid cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hee Chul Park, Professor, Study Chair — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thermo-radio-chemotherapy Arm
Started | 14
Completed | 13
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Thermo-radio-chemotherapy Arm
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants] — age, categorical (years)
  Participants
    <=18 years | 0
    Between 18 and 65 years | 8
    >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 60 [32 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 14

OUTCOME MEASURES:

1. Primary Outcome: Curative Resection Rate of Laparoscopic TME
Description: Curative resection rate of laparoscopic TME after CCRT and hyperthermia treament
Time Frame: expected average of 6 weeks after neoadjuvant treatement
Measure: Count of Participants; unit: Participants
Arm/Group | Thermo-radio-chemotherapy Arm
Number analyzed (Participants) | 10
Participants | 9

2. Primary Outcome: Pathologic Response of Thermo-radio-chemotherapy
Description: The pathologic response was assessed according to the Dworak's system. The pathologic response grades were as follows: grade 0, no response; grade 1, dominant tumor mass with obvious fibrosis, vasculopathy, or both (minimal response); grade 2, dominant fibrotic changes with a few easy-to-find tumor cells or groups (moderate response); grade 3, few (difficult to find microscopically) tumor cells in fibrotic tissue with or without mucous substance (near complete response); and grade 4, no viable tumor (complete response)
Time Frame: expected average of 6 weeks after neoadjuvant treatement
Population: 40% of pathologic response rate of laparoscopic TME after CCRT and hyperthermia treament
Measure: Number; unit: participants
Arm/Group | Thermo-radio-chemotherapy Arm
Number analyzed (Participants) | 10
participants | 4

3. Primary Outcome: Adverse Event of Laparoscopic TME and Hyperthermia With CCRT
Description: Adverse event according to CTCAE V 4.0 after laparoscopic TME and hyperthermia with CCRT
Time Frame: expected average of 16 weeks after neoadjuvant treatement
Measure: Count of Participants; unit: Participants
Arm/Group | Thermo-radio-chemotherapy Arm
Number analyzed (Participants) | 10
Participants | 0

4. Secondary Outcome: Rate of Open TME
Description: Rate of open TME was measured as ten percent
Time Frame: expected average of 6 weeks after neoadjuvant treatement
Measure: Number; unit: participants
Groups:
- Thermo-radio-chemotherapy Arm: Radiation: Hyperthermia with concurrent chemo-radiation therapy
Arm/Group | Thermo-radio-chemotherapy Arm
Number analyzed (Participants) | 10
participants | 1

5. Secondary Outcome: Pathologic Complete Response of Hyperthermia With CCRT
Description: Pathologic complete response of hyperthermia with CCRT was achieved in 20% of participants
Time Frame: expected average of 6 weeks after neoadjuvant treatement
Measure: Number; unit: participants
Arm/Group | Thermo-radio-chemotherapy Arm
Number analyzed (Participants) | 10
participants | 2

ADVERSE EVENTS:
Time Frame: expected average of 16 weeks after neoadjuvant treatement
Arm/Group | Thermo-radio-chemotherapy Arm
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes